CLINICAL TRIAL: NCT06044142
Title: Photodynamic Therapy by Curcumin VS Photo-bio-modulation Therapy of Oral Mucositis in Pedology Patient Undergoing Anti-Cancer Non-invasive Treatment
Brief Title: Curcumin VS Photo-bio-modulation Therapy of Oral Mucositis in Pediatric Patients Undergoing Anti-Cancer Non-invasive Treatment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Riyadh Elm University (Other)
Responsible Party: Principal Investigator, Tayyaba Zeeshan, Associate Professor, Director of Oral Diagnosis Postgraduate Program, Riyadh Elm University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FRP/2023/519/1030
Record Dates: First submitted 2023-09-05; First posted 2023-09-21 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-08

CONDITIONS: Oral Mucositis; Pediatric Cancer
Keywords: Curcumin; Photodynamic therapy; Pedology; Photo-bio-modulation; Oral Mucositis
MeSH Terms: conditions — Stomatitis; Neoplasms | interventions — Curcumin; Lasers

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A: Oral Mucositis (Experimental): Group A will be submitted to photodynamic therapy (Curcumin and red laser, λ450 nm) with 142 J/cm2, 100mW. The number of points will be calculated based on the size of lesion (1 laser shot per cm2 of lesion). The intervention will be repeated daily until cure of the oral mucositis was attained.
  Interventions: Drug: Curcumin; Device: Laser
- Group B: Oral Mucositis (Placebo Comparator): Group B (control group) will be submitted to low level (LL) laser therapy (λ660 nm) with 1J energy per point at 100mW power output for 10 seconds on daily basis until the lesion is clinically cured. The light will be applied perpendicular to the lesion on a continuous mode. The number of points will be calculated similarly as mentioned for patients included in Group A.
  Interventions: Device: Laser

INTERVENTIONS:
Drug: Curcumin — Curcumin and low laser therapy will be used on patients undergoing chemotherapy
  Arms: Group A: Oral Mucositis
Device: Laser — Low level laser therapy

SUMMARY:
The main objective of this study is to assess the impact of non-invasive photodynamic therapy by Curcumin and photo-bio-modulation low level (LL) laser treatment in managing mucositis induced by chemotherapy in pediatric patients.

A randomized clinical trial will be conducted involving 90 patients aged between 3 years and 15 years. The trial will be open, controlled, and blinded, and the patients will be divided into two groups.

DETAILED DESCRIPTION:
The study will be designed based on the Consolidated Standards of Reporting Trials (CONSORT) and conducted on approval from the Ethics Committee of the University. It will be a randomized controlled trial conducted among 90 pediatric patients of 3 years to 15 years age group. The inclusion criterion for the study will be i) patients in age group of 3 years to 15 years and ii) mucositis (categorized >1) based on the guidelines of WHO Toxicity Criteria. Pediatric patients having a malignant type of neoplasm and/or clinically evident oral microbial disease and/or with serious medical issues will be excluded from the study.

The oral mucositis will be diagnosed by a dentist available at the site of tertiary care hospital for chemotherapy. The potential participant will be referred to the research group for inclusion in the study based on the defined inclusion criterion. The procedure of research will be explained to the guardians of the participants. On acceptance, the guardians will be requested to sign the informed consent form.

The patients will considered as a new case for intervention on commencement of each chemo-therapy cycle. The patients will again added to a new randomized controlled trial if encountered an episode of oral mucositis.

Intervention for Photodynamic and Laser Therapy Prior to intervention of laser and photodynamic therapy the patients will be educated and instructed to maintain oral hygiene during cancer treatments. The instructions included brushing teeth with adequate amount of toothpaste and record it on follow-up chart. Later on inspection by the research team, if a patient is diagnosed with any carious lesion, retained root or gingival infection associated with dental plaque will be categorized as excluded from study. The procedure will be performed at beside for the patients admitted in the hospital; whereas outpatients will be seated on dental chairs of outpatient clinics.

An open controlled and blind, randomized clinical trial will be conducted with 45 patients, from 3 years to 15 years old, who will be divided into two groups. Group A will be submitted to photodynamic therapy (Curcumin and red laser, λ450 nm) with 142 J/cm2, 100mW. The number of points will be calculated based on the size of lesion (1 laser shot per cm2 of lesion). The intervention will be repeated daily until cure of the oral mucositis was attained. The clinical cure will be categorized as restoring the normal physiological functions such as chewing, swallowing and phonation without any symptoms of pain; additionally signs of tissue regeneration are evident.

Group B (control group) will be submitted to low level (LL) laser therapy (λ660 nm) with 1J energy per point at 100mW power output for 10 seconds on daily basis until the lesion was clinically cured. The light will be applied perpendicular to the lesion on a continuous mode. The number of points will calculated similarly as mentioned for patients included in Group A.

Oral Mucositis Evaluation After inter-examiner reliability test, the patients will be evaluated by the by the research group. The scale proposed and accepted by World Health Organization (WHO) will be used to categorize the changes in oral mucositis condition evaluated over time in four different categories: i) Category 0 = Absence of change in condition; ii) Category I = Persistence of erythematous condition and failure to have solid food; iii) Category II = Persistence of erythematous condition with solid dietary food intake iv) Category III: Presence of painful erythematous lesion with liquids as a dietary intake; and Category IV: patient with special mode for dietary intake (parenteral or enteral).

For evaluating the intensity of paint and variation in function, the ChIME scale will be used. The data will be recorded on special designed forms. The patients will be divided randomly and later treated with lasers and photodynamic therapy.

ELIGIBILITY:
Inclusion Criteria:

* patients in age group of 3 years to 15 years
* mucositis (categorized >1) based on the guidelines of WHO Toxicity Criteria
* must be able to open the mouth properly

Exclusion Criteria:

* Patients with age less than 3 years and more than 15 years of age
* patients with systemic diseases

Ages: 3 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
Assess the impact of non-invasive photodynamic therapy by Curcumin | 5 months
  The scale proposed and accepted by World Health Organization (WHO) will be used to categorize the changes in oral mucositis condition evaluated over time in four different categories: i) Category 0 = Absence of change in condition; ii) Category I = Persistence of erythematous condition and failure to have solid food; iii) Category II = Persistence of erythematous condition with solid dietary food intake iv) Category III: Presence of painful erythematous lesion with liquids as a dietary intake; and Category IV: patient with special mode for dietary intake (parenteral or enteral).
  For evaluating the intensity of paint and variation in function, the ChIME scale will be used. The data will be recorded on special designed forms.
Assess the impact of photo-bio-modulation low level (LL) laser treatment in managing mucositis | 5 months
  The scale proposed and accepted by World Health Organization (WHO) will be used to categorize the changes in oral mucositis condition evaluated over time in four different categories: i) Category 0 = Absence of change in condition; ii) Category I = Persistence of erythematous condition and failure to have solid food; iii) Category II = Persistence of erythematous condition with solid dietary food intake iv) Category III: Presence of painful erythematous lesion with liquids as a dietary intake; and Category IV: patient with special mode for dietary intake (parenteral or enteral).
  For evaluating the intensity of paint and variation in function, the ChIME scale will be used. The data will be recorded on special designed forms.

CONTACTS AND LOCATIONS:
Locations (1):
- Riyadh Elm University, Riyadh, Ar Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided